CLINICAL TRIAL: NCT04336228
Title: The Role of Serotonin in Compulsive Behavior in Humans: Underlying Brain Mechanisms
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Cambridge (Other); Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Gitte Moos Knudsen, Professor, MD, DMSc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-18038325
Record Dates: First submitted 2020-03-25; First posted 2020-04-07 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Obsessive-Compulsive Disorder/High Compulsive Individuals; Healthy Individuals
Keywords: Serotonin; Cognition; Emotion; Neural Activation
MeSH Terms: interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy Control Group (Placebo Comparator): The healthy placebo control group will be administered the exact same procedure as the intervention group, the only difference being that this group will be administered a placebo tablet.
  Interventions: Drug: Placebo oral tablet
- Obsessive-Compulsive Disorder / High Compulsivity Control Group (Placebo Comparator): The OCD/high compulsivity placebo control group will be administered the exact same procedure as the intervention group, the only difference being that this group will be administered a placebo tablet.
  Interventions: Drug: Placebo oral tablet
- Healthy Intervention Group (Experimental): The healthy intervention group will be administered 20mg of Escitalopram daily for 3-4 weeks.
  Interventions: Drug: Escitalopram
- Obsessive-Compulsive Disorder / High Compulsivity Intervention Group (Experimental): The OCD/high compulsivity intervention group will be administered 20mg of Escitalopram daily for 3-4 weeks.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — 20mg daily for 3-4 weeks.
  Other Names: Escitalopram STADA
  Arms: Healthy Intervention Group; Obsessive-Compulsive Disorder / High Compulsivity Intervention Group
Drug: Placebo oral tablet — 20mg placebo tablet daily for 3-4 weeks.
  Other Names: calcium tables
  Arms: Healthy Control Group; Obsessive-Compulsive Disorder / High Compulsivity Control Group

SUMMARY:
The aim of this project is to investigate:

* The status of the central serotonin (5-hydroxytryptamine, 5-HT) system in compulsive behaviour and how it is affected by sub-chronic escitalopram administration
* The mechanisms underlying how sub-chronic administration of escitalopram affects the central 5-HT system
* How changes in cognitive performance, including the balance between habitual and goal-directed mechanisms, are affected in compulsive behaviour by boosting 5-HT function
* How functional brain changes in cognitive function measured with magnetic resonance imaging relate to altered 5-HT function following escitalopram administration.

DETAILED DESCRIPTION:
Previous studies have shown that 5-HT is strongly implicated in compulsive behaviours in experimental animals. Manipulation of 5-HT influences neuronal interactions underlying action selection. Reduced forebrain 5-HT causes perseveration and impairs goal-directed behaviour under reward but not punishment. Dysfunctional 5-HT neurotransmission has also been implicated in Obsessive-Compulsive Disorder (OCD) based on the selective efficacy of relatively high doses of selective serotonin reuptake inhibitors (SSRIs) in treating this disorder. Hitherto, it is unknown whether there is a primary defect in the serotonergic system or whether SSRIs ameliorate symptoms by modulating other brain neurotransmitter pathways. So far, only one study of central 5-HT release in OCD patients has been conducted and its methodology may be questioned.

A number of behavioural and cognitive features of OCD, including endophenotype markers that appear to characterise the disorder have been determined. These include a shift in cognitive control from a goal-directed strategy to a habitual (stimulus-response, S-R) strategy, cognitive rigidity in terms of both reversal learning and attentional set-shifting, impaired response inhibition and planning, and a tendency to over-respond to spurious negative feedback in a probabilistic learning paradigm. Neural substrates of these deficits are being investigated using brain imaging methodologies based on magnetic resonance and preliminary evidence suggests an over-active medial prefrontal cortex-caudate nucleus circuits and underactive lateral prefrontal cortex-putamen circuits. However, little evidence exists that relates to the hypothesis of an over-active habit system in this disorder or to the role of serotonin in all these cognitive and behavioural deficits observed in OCD and compulsivity in general.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with high scores on obsessive-compulsive traits (with or without a diagnosis of OCD established by a psychiatrist) and healthy volunteers (male or female) between 18 and 70 years. Compulsive individuals without an OCD diagnosis are individuals without a history of psychiatric or other major medical conditions but scoring abnormally high on the Obsessive-Compulsive Inventory (OCI) questionnaire.

Exclusion Criteria:

* Current or previous neurological disease, severe somatic disease, or consumption of medical drugs likely to influence the test results
* Non- fluent in Danish or pronounced visual or auditory impairments
* Current or past learning disability.
* Pregnancy
* Lactation
* Participation in experiments with radioactivity (> 10 mSv) within the last year or significant occupational exposure to radioactivity.
* Contraindications for MRI (pacemaker, metal implants, etc.).
* Allergy to the ingredients in the administered drug.
* Abnormal ECG (e.g. prolonged QT syndrome).
* Dizzy when changing from supine to upright position (e.g. postural orthostatic tachycardia syndrome).
* Mild hypotension (blood pressure below 100/70 mmHg) or hypertension (blood pressure above 140/90 mmHg).
* Head injury or concussion resulting in loss of consciousness for more than 2 min.
* Alcohol or drug abuse
* Drug use other than tobacco and alcohol within the last 30 days.
* Hash > 50 x lifetime.
* Drugs > 10 x lifetime (for each substance).
* Current medication with serotonergic acting compounds. Use of other psychoactive substances must be stable at least one month prior to inclusion and maintained throughout the study.
* Severe physical impairments affecting eyesight or motor performance.
* For the OCD group: other Axis I mental disorder as primary diagnosis according to ICD-10 criteria.
* For healthy volunteers: any current or former primary psychiatric disorder (Axis I WHO ICD-10 diagnostic classification).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Learning Primary Outcome 1 measured with Probability Reversal Learning test: Mean errors Stage 1 (Learning) | 3 years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Primary Outcome 2 measured with Probability Reversal Learning test: Mean errors Stage 2 (Reversal) | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Primary Outcome 3 measured with Deterministic Reversal Learning test: Percent correct per stage | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Inhibition Primary Outcome 1 measured with Interleaved Stop Signal Task/Go-NoGo: Stop Signal Reaction Time | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Flexibility Primary Outcome 1 measured with 3Dimensional Intra/Extra Dimensional Shift test: Extra Dimensional Set Errors | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Flexibility Primary Outcome 2 measured with Sequential model-based model-free test: Model-based Model-free Weight | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Social Cognition Primary Outcome 1 measured with EMOTICOM Moral Emotions Task: Agent Guilt Score | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Social Cognition Primary Outcome 2 measured with EMOTICOM Moral Emotions Task: Agent Shame Score | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. The false discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Primary Outcome 1 measures with EMOTICOM Intensity Morphing: Affective bias in decreasing condition | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Primary Outcome 2 measured with EMOTICOM Emotion Recognition Task: Affective bias for D' | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Primary Outcome 3 measured with EMOTICOM Intensity Morphing task: Detection threshold decreasing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Primary Outcome 4 measured with EMOTICOM Emotion Recognition task: D'Prime for emotion recognition | 3 Years
  Emotion Recognition Task. Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Memory Primary Outcome 1 measured with CANTAB Paired Associates Learning: Total Errors Adj | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Biofluids | 3 Years
  Serum Escitalopram levels
Positron emission tomography (PET) Imaging: Cerebral [11C]SB207145 PET binding. | 3 Years
  Collected before and after participant's intervention.
Neural Activations and Correlations measured with functional magnetic resonance imaging (fMRI) paradigm named Slip of Actions | 3 Years
  Imaging outcomes will be Family-Wise Error (FWE) corrected using Random Field Theory as implemented in SPM12.
Neural Activations and Correlations measured with functional magnetic resonance imaging (fMRI) paradigm named Cohabit | 3 Years
  Imaging outcomes will be Family-Wise Error (FWE) corrected using Random Field Theory as implemented in SPM12Co-habit fMRI paradigm Imaging outcomes will be FWE corrected using Random Field Theory as implemented in SPM12.
Neural Activations and Correlations measured with functional magnetic resonance imaging (fMRI) paradigm named Faces | 3 Years
  Imaging outcomes will be Family-Wise Error (FWE) corrected using Random Field Theory as implemented in SPM12.
Resting State fMRI | 3 Years
  Imaging outcomes will be Family-Wise Error (FWE) corrected using Random Field Theory as implemented in SPM12.
Structural Voxel-based morphometry (VBM) MRI | 3 Years
  Imaging outcomes will be Family-Wise Error (FWE) corrected using Random Field Theory as implemented in SPM12.
Diffusion Tensor Imaging MRI | 3 Years
Habit formation outcome 1: response times for each day of training | 3 Years
  Daily app training paradigm
Habit formation outcome 2: mean errors per sequence and moves | 3 Years
  Daily app training paradigm
Habit formation outcome 3: confidence and enjoyable rates. | 3 Years
  Daily app training paradigm

SECONDARY OUTCOMES:
Learning Secondary Outcome 1 measured with Probability Reversal Learning test: Stage 1 Reward-Stay/Lose-Shift behaviour | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Secondary Outcome 2 measured with Probability Reversal Learning test: Stage 1 Reward/Punishment learning | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Secondary Outcome 3 measured with Probability Reversal Learning test: Stage 1. Stimulus Stickiness | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Secondary Outcome 4 measured with Probability Reversal Learning test: Stage 2 Reward-Stay/ Lose-Shift behaviour | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Secondary Outcome 5 measured with Probability Reversal Learning test: Stage 2 Reward/Punishment learning | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Secondary Outcome 6 measured with Probability Reversal Learning test: Stage 2. Stimulus Stickiness | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Learning Secondary Outcome 7 measured with Deterministic Reversal Learning test: Reward-Stay/ Lose-Shift behaviour | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Flexibility Secondary Outcome 1 measured with Sequential Model-Based/Model-Free test: Proportion of Stays | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Flexibility Secondary Outcome 2 measured with Sequential Model-Based/Model-Free test: Exploration | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Flexibility Secondary Outcome 3 measured with Sequential Model-Based/Model-Free test: Stimulus Stickiness | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Flexibility Secondary Outcome 4 measured with Sequential Model-Based/Model-Free test: Learning rate | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Flexibility Secondary Outcome 5 measured with 3Dimensional Intra/Extra Dimensional Shift test: Pre Extra Dimension Set Errors | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Flexibility Secondary Outcome 6 measured with 3Dimensional Intra/Extra Dimensional Shift test: Latency | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Inhibition Secondary Outcome 1 measured with Interleaved Stop Signal Task/Go-NoGo: Go reaction time | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Inhibition Secondary Outcome 2 measured with Interleaved Stop Signal Task/Go-NoGo: Go omission error rate | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Inhibition Secondary Outcome 3 measured with Interleaved Stop Signal Task/Go-NoGo: Go commission error rate | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Inhibition Secondary Outcome 4 measured with Interleaved Stop Signal Task/Go-NoGo: No-Go error rate | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Executive Function Secondary Outcome 1 measured with 3Dimensional Intra/Extra Dimensional Shift test: Total Errors Adjusted | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Secondary Outcome 1 measured with EMOTICOM Intensity Morphing Task: Detection threshold increasing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Secondary Outcome 2 measured with EMOTICOM Intensity Morphing Task: Affective bias in increasing condition | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Secondary Outcome 3 measured with EMOTICOM Emotion Recognition Task: Affective bias for Hit Rate | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Emotion Recognition Secondary Outcome 4 measured with EMOTICOM Emotion Recognition Task.: Hit Rate for Emotion Recognition | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Faces and geometric figure discrimination Outcome 1 measured with fMRI faces paradigm: Accuracy | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Behavioural outcomes with Faces and geometric figure discrimination Outcome 2 measured with fMRI faces paradigm: Response Speed | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Behavioural outcomes with fMRI paradigm slip of Actions : accuracy and latency | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Behavioural outcomes with fMRI paradigm Co-habit: accuracy and latency. | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Memory Outcome 1 measured with CANTAB Paired Associates Learning test: First Trial Memory Score | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Memory Outcome 2 measured with Letter-number sequencing test: Total score | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Memory Primary outcome 3 measured with Verbal Affective Memory Test-26: Latent variable model of the association between positive, negative and neutral word recall and 5-HT4R binding | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Risky Decision Making Outcome Outcome 1 measured with EMOTICOM Cambridge Gamble Task: Quality of Decision Making | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Risky Decision Making Outcome 2 measured with EMOTICOM Cambridge Gamble Task: Risk Adjustment | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Risky Decision Making Outcome 3 measured with EMOTICOM Cambridge Gamble Task: Overall Proportion Bet | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Risky Decision Making Outcome 4 measured with EMOTICOM Cambridge Gamble Task: Deliberation Time | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Psychomotor Speed Outcome 1 measured with CANTAB Reaction Time Task: Simple reaction time | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain.
Intelligence Quotient (IQ) outcome 1 measured with Reynolds Intellectual assessment Scales subtest "guess what" and "what does not fit": Total age adjusted score | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains. False discovery rate (FDR) correction, for multiple comparisons, using the Benjamini-Hochberg procedure will be applied to the outcomes within each cognitive domain
Interpersonal Reactivity Index (IRI) Score | 3 Years
Obsessive- Compulsive Inventory (OCI)- state Score | 3 Years
Obsessive- Compulsive Inventory- trait Score | 3 Years
Brief Symptom Inventory (BSI) Score | 3 Years
Pittsburgh Sleep Quality Index Score | 3 Years
Profile of Mood State Score | 3 Years
Beck Depression Inventory-II Score | 3 Years
  Contain 21-items, scored on a scale value of 0 to 3
State-Trait Anxiety Inventory Scale Score | 3 Years
  Contain 40-items
State and Trait Aggression Questionnaire Score | 3 Years
Barratt Impulsiveness Scale-State Score | 3 Years
Visual Analogue Scale Score | 3 Years

OTHER OUTCOMES:
Emotion Recognition Other Outcome 1: Detection threshold decreasing Happy - Intensity Morphing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 2: Detection threshold decreasing Sad - Intensity Morphing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 3: Detection threshold decreasing Anger - Intensity Morphing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 4: Detection threshold decreasing Fear - Intensity Morphing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 5: Detection threshold decreasing Disgust - Intensity Morphing | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 6: D' Happy - Emotion Recognition Task | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 7: D' Sad - Emotion Recognition Task | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 8: D' Fear - Emotion Recognition Task | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Emotion Recognition Other Outcome 9: D' Anger - Emotion Recognition Task | 3 Years
  Outcome variables have been grouped a priori into carefully defined cognitive domains.
Activity Level Score | 3 Years
Behavioural Inhibition/ Behavioural Avoidance Scale Score | 3 Years
The Compulsive Personality Assessment Scale Score | 3 Years
Sexuality Questionnaire Score | 3 Years
Edinburgh Handedness Inventory Score | 3 Years
Revised NEO Personality Questionnaire Score | 3 Years
Family History Assessment Module Score | 3 Years
Positive Life Events Score | 3 Years
Stressful Life Events Score | 3 Years
Perceived stress scale | 3 Years
Barratt Impulsiveness Scale-Trait Score | 3 Years
The Penn State Worry Questionnaire- Trait Score | 3 Years
The Penn State Worry Questionnaire- State Score | 3 Years
The Self-Control Scale- Trait Score | 3 Years
The Self-Control Scale- State Score | 3 Years
State- Trait Anxiety Inventory- Trait Score | 3 Years
The Warwick-Edinburgh Mental Well-being Scale -State Score | 3 Years
The Warwick-Edinburgh Mental Well-being Scale -Trait Score | 3 Years
Mindful Attention and Awareness Scale -State Score | 3 Years
Mindful Attention and Awareness Scale -Trait Score | 3 Years
The Intolerance of Uncertainty Scale - Trait Score | 3 Years
The Intolerance of Uncertainty Scale - State Score | 3 Years
Verran and Snyder-Halpern (VSH) Sleep Scale Score | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Gitte M. Knudsen, Professor, Study Chair — Neurobiology Research Unit, Rigshospitalet
Locations (1):
- Neurobiology Research Unit, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study all data will be uploaded to the existing Center for Integrated Molecular Brain Imaging (CIMBI) Database. Researchers may apply for access to the data.
Time Frame: Upon completion of the study.
Access Criteria: Researchers may apply for access to the data.
URL: https://nru.dk/index.php/research-menu/research-groups/115-the-cimbi-database-and-biobank

REFERENCES:
- [Background] Clarke HF, Dalley JW, Crofts HS, Robbins TW, Roberts AC. Cognitive inflexibility after prefrontal serotonin depletion. Science. 2004 May 7;304(5672):878-80. doi: 10.1126/science.1094987. PMID 15131308
- [Background] Dayan P, Huys QJ. Serotonin in affective control. Annu Rev Neurosci. 2009;32:95-126. doi: 10.1146/annurev.neuro.051508.135607. PMID 19400722
- [Background] Palminteri S, Clair AH, Mallet L, Pessiglione M. Similar improvement of reward and punishment learning by serotonin reuptake inhibitors in obsessive-compulsive disorder. Biol Psychiatry. 2012 Aug 1;72(3):244-50. doi: 10.1016/j.biopsych.2011.12.028. Epub 2012 Feb 10. PMID 22325972
- [Background] Pelloux Y, Dilleen R, Economidou D, Theobald D, Everitt BJ. Reduced forebrain serotonin transmission is causally involved in the development of compulsive cocaine seeking in rats. Neuropsychopharmacology. 2012 Oct;37(11):2505-14. doi: 10.1038/npp.2012.111. Epub 2012 Jul 4. PMID 22763621
- [Background] Groman SM, James AS, Seu E, Crawford MA, Harpster SN, Jentsch JD. Monoamine levels within the orbitofrontal cortex and putamen interact to predict reversal learning performance. Biol Psychiatry. 2013 Apr 15;73(8):756-62. doi: 10.1016/j.biopsych.2012.12.002. Epub 2013 Jan 16. PMID 23332512
- [Background] Worbe Y, Palminteri S, Savulich G, Daw ND, Fernandez-Egea E, Robbins TW, Voon V. Valence-dependent influence of serotonin depletion on model-based choice strategy. Mol Psychiatry. 2016 May;21(5):624-9. doi: 10.1038/mp.2015.46. Epub 2015 Apr 14. PMID 25869808
- [Background] el Mansari M, Bouchard C, Blier P. Alteration of serotonin release in the guinea pig orbito-frontal cortex by selective serotonin reuptake inhibitors. Relevance to treatment of obsessive-compulsive disorder. Neuropsychopharmacology. 1995 Oct;13(2):117-27. doi: 10.1016/0893-133X(95)00045-F. PMID 8597523
- [Background] Lissemore JI, Sookman D, Gravel P, Berney A, Barsoum A, Diksic M, Nordahl TE, Pinard G, Sibon I, Cottraux J, Leyton M, Benkelfat C. Brain serotonin synthesis capacity in obsessive-compulsive disorder: effects of cognitive behavioral therapy and sertraline. Transl Psychiatry. 2018 Apr 18;8(1):82. doi: 10.1038/s41398-018-0128-4. PMID 29666372
- [Background] Banca P, Voon V, Vestergaard MD, Philipiak G, Almeida I, Pocinho F, Relvas J, Castelo-Branco M. Imbalance in habitual versus goal directed neural systems during symptom provocation in obsessive-compulsive disorder. Brain. 2015 Mar;138(Pt 3):798-811. doi: 10.1093/brain/awu379. Epub 2015 Jan 6. PMID 25567322
- [Background] Gillan CM, Papmeyer M, Morein-Zamir S, Sahakian BJ, Fineberg NA, Robbins TW, de Wit S. Disruption in the balance between goal-directed behavior and habit learning in obsessive-compulsive disorder. Am J Psychiatry. 2011 Jul;168(7):718-26. doi: 10.1176/appi.ajp.2011.10071062. Epub 2011 May 15. PMID 21572165
- [Background] Apergis-Schoute AM, Gillan CM, Fineberg NA, Fernandez-Egea E, Sahakian BJ, Robbins TW. Neural basis of impaired safety signaling in Obsessive Compulsive Disorder. Proc Natl Acad Sci U S A. 2017 Mar 21;114(12):3216-3221. doi: 10.1073/pnas.1609194114. Epub 2017 Mar 6. PMID 28265059
- [Background] Chamberlain SR, Fineberg NA, Blackwell AD, Robbins TW, Sahakian BJ. Motor inhibition and cognitive flexibility in obsessive-compulsive disorder and trichotillomania. Am J Psychiatry. 2006 Jul;163(7):1282-4. doi: 10.1176/ajp.2006.163.7.1282. PMID 16816237
- [Background] Chamberlain SR, Fineberg NA, Menzies LA, Blackwell AD, Bullmore ET, Robbins TW, Sahakian BJ. Impaired cognitive flexibility and motor inhibition in unaffected first-degree relatives of patients with obsessive-compulsive disorder. Am J Psychiatry. 2007 Feb;164(2):335-8. doi: 10.1176/ajp.2007.164.2.335. PMID 17267798
- [Background] Vaghi MM, Vertes PE, Kitzbichler MG, Apergis-Schoute AM, van der Flier FE, Fineberg NA, Sule A, Zaman R, Voon V, Kundu P, Bullmore ET, Robbins TW. Specific Frontostriatal Circuits for Impaired Cognitive Flexibility and Goal-Directed Planning in Obsessive-Compulsive Disorder: Evidence From Resting-State Functional Connectivity. Biol Psychiatry. 2017 Apr 15;81(8):708-717. doi: 10.1016/j.biopsych.2016.08.009. Epub 2016 Aug 11. PMID 27769568
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Delgado P, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. II. Validity. Arch Gen Psychiatry. 1989 Nov;46(11):1012-6. doi: 10.1001/archpsyc.1989.01810110054008. PMID 2510699
- [Background] Haahr ME, Fisher PM, Jensen CG, Frokjaer VG, Mahon BM, Madsen K, Baare WF, Lehel S, Norremolle A, Rabiner EA, Knudsen GM. Central 5-HT4 receptor binding as biomarker of serotonergic tonus in humans: a [11C]SB207145 PET study. Mol Psychiatry. 2014 Apr;19(4):427-32. doi: 10.1038/mp.2013.147. Epub 2013 Nov 5. PMID 24189342
- [Background] Foa, E. B. et al. The validation of a new obsessive-compulsive disorder scale: The obsessive-compulsive inventory. Psychological Assessment 10(3), 206-214, 1998.

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT04336228/SAP_000.pdf